CLINICAL TRIAL: NCT06477289
Title: Peripheral Arterial Tonometry and Neurocognition in Sickle Cell Disease
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PATSCANS
Record Dates: First submitted 2024-06-20; First posted 2024-06-27 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will examine sleep disordered breathing and sleep quality in participants (ages 12-18) diagnosed with sickle cell disease of any genotype. We will utilize remote peripheral arterial tonometry (PAT) and questionnaires to evaluate difficulties with sleep. PAT assessments will occur remotely in the homes of participants.

Neurocognitive, behavioral, and neuroimaging evaluations will occur on the same day as a routine clinic visit.

Primary Objective:

Evaluate the relationship between nocturnal oxyhemoglobin saturation (SpO2) and neurocognitive functioning (working memory and verbal comprehension) in children (ages 12-18) diagnosed with sickle cell disease controlling for age, genotype, and social vulnerability.

Secondary Objective:

Assess differences in white matter integrity, silent cerebral infarcts, neuroinflammation, and functional connectivity among children (ages 12-18) diagnosed with sickle cell disease with and without sleep disordered breathing after controlling for age.

Assess differences in self- and caregiver-reported mood and pain severity among children (ages 12-18) diagnosed with sickle cell disease with and without sleep disordered breathing after controlling for age.

Exploratory Objectives:

Explore the relationship between nocturnal oxyhemoglobin saturation (SpO2) and neurocognitive functioning (attention, processing speed, verbal memory, visual memory, motor dexterity) in children (ages 12-18) diagnosed with sickle cell disease controlling for age, genotype, and social vulnerability.

Assess the feasibility of an ultraportable ring oximeter (BodimetricsCircul+ Ring) in children (ages 12-18) diagnosed with sickle cell disease.

Assess the concordance between the Circul+Ring with the WatchPAT in children (ages 12-18) diagnosed with sickle cell disease.

DETAILED DESCRIPTION:
Interested participants will be consented in-person or virtually. Consented participants will be mailed the equipment (WatchPAT and Circul+ Ring) to conduct the remote assessment. Additional questionnaires will also be sent via mail or email for the participant to complete prior to collecting data on sleep behaviors. After receiving the questionnaires and equipment, a virtual session will be conducted with the participant to provide education on how to use the equipment and complete the included questionnaires. Participants will wear the WatchPAT and Circul+ Ring overnight for three days and data will be captured remotely. After wearing the devices for three consecutive nights, the participant will attend a research visit within approximately the next two weeks where they will complete performance based neurocognitive assessments, behavioral rating forms, and neuroimaging.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with sickle cell disease of any genotype
* Participant in the Sickle Cell Clinical Research and Intervention Program
* Between 12-18 years of age at the time of enrollment
* English is the primary language
* Access to a smartphone or tablet for use with the Circul+ Ring

Exclusion Criteria:

* History of an intellectual disability
* History of a traumatic brain injury or seizure disorder
* History of a stroke
* Undergoing potential curative treatment for SCD (stem cell transplant or gene therapy)
* Currently prescribed an intervention for a sleep disorder
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Ages: 12 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study will recruit participants ages 12-18 diagnosed with sickle disease of any genotype.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the relationship between nocturnal oxyhemoglobin saturation (SpO2) and neurocognitive functioning (working memory and verbal comprehension) in children (ages 12-18) diagnosed with sickle cell disease. | Baseline remote sleep assessment over 3 days followed by in-clinic assessment.
  A linear regression model will be used to assess the relationship between SpO2 and neurocognitive functioning after adjusting for age, genotype, and social vulnerability.

SECONDARY OUTCOMES:
Assess differences in white matter integrity among children (ages 12-18) diagnosed with sickle cell disease with and without sleep disordered breathing. | Baseline remote sleep assessment over 3 days followed by in-clinic assessment.
  This study will measure resting-state BOLD signal in SCD patients after assessing nocturnal oxyhemoglobin saturation. The primary endpoint is the whole brain BOLD response and functional connectivity among brain regions within the default mode, fronto-parietal, executive control, salience, sensorimotor, and other resting state networks. Then we will compare differences in white matter integrity based on the structural connectivity connectome for the working memory network, silent cerebral infarcts, neuroinflammation, and functional connectivity among children with and without sleep disordered breathing.
Assess differences in silent cerebral infarcts among children (ages 12-18) diagnosed with sickle cell disease with and without sleep disordered breathing. | Baseline remote sleep assessment over 3 days followed by in-clinic assessment.
  This study will measure resting-state BOLD signal in SCD patients after assessing nocturnal oxyhemoglobin saturation. The primary endpoint is the whole brain BOLD response and functional connectivity among brain regions within the default mode, fronto-parietal, executive control, salience, sensorimotor, and other resting state networks. Then we will compare differences in white matter integrity based on the structural connectivity connectome for the working memory network, silent cerebral infarcts, neuroinflammation, and functional connectivity among children with and without sleep disordered breathing.
Assess differences in neuroinflammation, among children (ages 12-18) diagnosed with sickle cell disease with and without sleep disordered breathing. | Baseline remote sleep assessment over 3 days followed by in-clinic assessment.
  This study will measure resting-state BOLD signal in SCD patients after assessing nocturnal oxyhemoglobin saturation. The primary endpoint is the whole brain BOLD response and functional connectivity among brain regions within the default mode, fronto-parietal, executive control, salience, sensorimotor, and other resting state networks. Then we will compare differences in white matter integrity based on the structural connectivity connectome for the working memory network, silent cerebral infarcts, neuroinflammation, and functional connectivity among children with and without sleep disordered breathing.
Assess differences in functional connectivity among children (ages 12-18) diagnosed with sickle cell disease with and without sleep disordered breathing after controlling for age. | Baseline remote sleep assessment over 3 days followed by in-clinic assessment.
  This study will measure resting-state BOLD signal in SCD patients after assessing nocturnal oxyhemoglobin saturation. The primary endpoint is the whole brain BOLD response and functional connectivity among brain regions within the default mode, fronto-parietal, executive control, salience, sensorimotor, and other resting state networks. Then we will compare differences in white matter integrity based on the structural connectivity connectome for the working memory network, silent cerebral infarcts, neuroinflammation, and functional connectivity among children with and without sleep disordered breathing.
Assess differences in self- and caregiver-reported mood and pain severity among children (ages 12-18) diagnosed with sickle cell disease with and without sleep disordered breathing after controlling for age. | Baseline remote sleep assessment over 3 days followed by in-clinic assessment.
  The general linear regression model is then used to assess the relationship of functional connectivity and to assess the relationship of self- and caregiver-reported mood and pain severity with sleep disordered breathing with controlling for age in the model. As a secondary analysis, we will also associate continuous obstructive and central AHI with functional connectivity and self- and caregiver-reported mood and pain severity using linear regression model with adjusting for age.

OTHER OUTCOMES:
Explore the relationship between nocturnal oxyhemoglobin saturation (SpO2) and neurocognitive functioning (attention, processing speed, verbal memory, visual memory, motor dexterity) in children (ages 12-18) diagnosed with sickle cell disease controlling | Baseline remote sleep assessment over 3 days followed by in-clinic assessment.
  A linear regression model will be used to assess the relationship between SpO2 and neurocognitive functioning after adjusting for age, genotype, and social vulnerability
Assess the feasibility of an ultraportable ring oximeter (BodimetricsCircul+ Ring) in children (ages 12-18) diagnosed with sickle cell disease. | Baseline remote sleep assessment over 3 days followed by in-clinic assessment.
  Feasibility of the Circul+Ring equipment will be defined as more than 50% of participants wearing Circul+Ring for at least one night's sleep. There is no power calculation needed for this feasibility objective. However, 55 participants give 92% power to detect a 20% difference at an assumed 70% of participants who will wear the ring for at least one night's sleep, with a significance level of 0.05 based on a one-sided test. The number of hours worn for the WatchPAT and Circul+Ring will be compared using Wilcoxon rank sum test. Descriptive statistics will be used to summarize the two-question survey.
Assess the concordance between the Circul+Ring with the WatchPAT in children (ages 12-18) diagnosed with sickle cell disease. | Baseline remote sleep assessment over 3 days followed by in-clinic assessment.
  To evaluate concordance, the nocturnal SpO2 obtained using the WatchPAT and a Circul+ Ring will be plotted against each other, and Pearson/Spearman correlations will be used to examine their relationship. The Bland-Altman method will be used to investigate the variability between the two measurements using the WatchPAT and Circul+ Ring. Lin's concordance correlation coefficient will be determined to demonstrate the level of agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Heitzer, Phd, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols